CLINICAL TRIAL: NCT00182481
Title: Long Term Management of Asthma (LOMA) Study- How Useful is the Sputum Count Compared With the Usual Clincal Variables?
Brief Title: LOMA: Long-Term Management of Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP#97-1549; MCT-44158
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2003-10

CONDITIONS: Asthma
Keywords: asthma treatment; induced sputum cell counts; asthma exacerbations; eosinophilic bronchitis; non-eosinophilic bronchitis
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Procedure: Induced sputum cell counts
Drug: inhaled corticosteroids and other asthma drugs

SUMMARY:
The purpose of this study was to determine whether the use of induced sputum cell counts could guide treatment of asthma more effectively than the use of symptoms and breathing tests. The main outcomes where the time to the first exacerbation and the number of exacerbations.

DETAILED DESCRIPTION:
Airway inflammation is an important component of asthma. It influences other components which include symptoms and airway functional (physiological) measurements. It is the primary target of treatment. However, it does not correlate closely with symptoms, need for symptomatic bronchodilator relief, or the physiological abnormalities. Furthermore, it can be of different types. As a result, physicians are poor at recognizing its presence or type. This is important because eosinophilic inflammation is responsive to corticosteroid while non-eosinophilic is not responsive.

The most comprehensive non-invasive or relatively non-invasive measurement of airway inflammation is by spontaneous or induced sputum cell counts. These are reliable, valid and responsive, the qualities of good measurements. They might therefore be clinically useful to guide individual treatment. In the present study we investigated this issue. We compared their use, in comparison with the use only of symptoms and spirometry, in preventing exacerbations of asthma. We chose prevention of exacerbations as the most important clinical outcome because these have the greatest impact on patient's quality of life, morbidity and healthcare utilization. The study comprised two Phases. In Phase 1, the minimum treatment to control sputum eosinophilia (as well as clinical criteria) in the Sputum Strategy, and clinical criteria in the Clinical Strategy, were established. In Phase 2, this minimum treatment was maintained and patients were seen every 3 momths and at exacerbations. The primary outcomes were the relative risk reduction for the occurrence of the first exacerbation and the length of time without exacerbation over 18-20 months in Phase 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. History of asthma for at least one year,confirmed objectively.
2. New or previously reviewed patients where the minimal treatment requirements have not been established within the last six months.

Exclusion Criteria:

1. Smokers or ex-smokers for less than 6 months with a smoking history of more than 10 pack years.
2. Other pulmonary co-morbidity (other than mild or moderate chronic airflow limitation).
3. Subjects having a co-existing illness that precludes them from the study.
4. Inability to give informed consent due to mental or legal reasons.
5. Pregnancy or lactation.
6. Known non-compliance with medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 1999-09; Study Completion 2001-09

PRIMARY OUTCOMES:
Relative risk reduction for the occurence of the first exacerbation and the length of time without exacerbation during Phase 2 of the study.

SECONDARY OUTCOMES:
Secondary outcomes were
The cellular type of exacerbation that was influenced,
The severity of asthma that was helped,
The dose of inhaled corticosteroid that was required,
Symptom control,
Quality of life,
FEV1
Methacholine PC20,
Exhaled NO,
Cost effectiveness and cost benefit of sputum cell counts, Airway structural changes
Skin bruising score.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Hargreave, MD, Principal Investigator — McMaster University; Louis-Philippe Boulet, MD, Principal Investigator — Laval University, Sainte-Foy, Quebec; Andre Cartier, MD, Principal Investigator — Hopital du Sacre Coeur, Montreal, PQ; Catherine Lemiere, MD, Principal Investigator — Hopital du Sacre Coeur, Montreal, PQ; Marcia Pizzichini, MD, Principal Investigator — Universidade Federal de Santa Catarina, Florianopolis, Brazil; Emilio Pizzichini, MD, Principal Investigator — Universidade Federal de Santa Catarina, Florianopolis, Brazil
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Cockcroft DW, Swystun VA. Asthma control versus asthma severity. J Allergy Clin Immunol. 1996 Dec;98(6 Pt 1):1016-8. doi: 10.1016/s0091-6749(96)80185-0. No abstract available. PMID 8977499
- [Background] Pavord ID, Brightling CE, Woltmann G, Wardlaw AJ. Non-eosinophilic corticosteroid unresponsive asthma. Lancet. 1999 Jun 26;353(9171):2213-4. doi: 10.1016/S0140-6736(99)01813-9. No abstract available. PMID 10392993
- [Background] Parameswaran K, Pizzichini E, Pizzichini MM, Hussack P, Efthimiadis A, Hargreave FE. Clinical judgement of airway inflammation versus sputum cell counts in patients with asthma. Eur Respir J. 2000 Mar;15(3):486-90. doi: 10.1034/j.1399-3003.2000.15.10.x. PMID 10759441
- [Background] Belda J, Leigh R, Parameswaran K, O'Byrne PM, Sears MR, Hargreave FE. Induced sputum cell counts in healthy adults. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):475-8. doi: 10.1164/ajrccm.161.2.9903097. PMID 10673188
- [Background] Gibson PG, Simpson JL, Saltos N. Heterogeneity of airway inflammation in persistent asthma : evidence of neutrophilic inflammation and increased sputum interleukin-8. Chest. 2001 May;119(5):1329-36. doi: 10.1378/chest.119.5.1329. PMID 11348936
- [Background] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Background] Djukanovic R, Sterk PJ, Fahy JV, Hargreave FE. Standardised methodology of sputum induction and processing. Eur Respir J Suppl. 2002 Sep;37:1s-2s. doi: 10.1183/09031936.02.00000102. No abstract available. PMID 12361359
- [Result] Pizzichini MMM, Jayaram L, Pizzichini E, Boulet LP, Lemière C, Efithmiades A, Cartier A, Hargreave FE. O exame das células no escarro induzido pode alterar as exacerbações da asma? O estudo LOMA. Respirtory Society Meeting. Bahia- Brazil. J Bras Pneum 2004, 30: S24
- [Result] Pizzichini MMM, Pizzichini E, Jayaram L, Boulet LP, Lemière C, Efithmiades A, Cartier A, Hargreave FE. Monitorando o tratamento da asma através do escarro induzido : efeito nas exacerbações. Latina America Thoracic Society Meeting, ALAT. Buenos Aires-Argentina. Arch de Bronconeumologia 2004, 40 S88-89.
- [Result] Jayaram L, Pizzichini MM, Cook RJ, Boulet LP, Lemiere C, Pizzichini E, Cartier A, Hussack P, Goldsmith CH, Laviolette M, Parameswaran K, Hargreave FE. Determining asthma treatment by monitoring sputum cell counts: effect on exacerbations. Eur Respir J. 2006 Mar;27(3):483-94. doi: 10.1183/09031936.06.00137704. PMID 16507847